CLINICAL TRIAL: NCT00623649
Title: A Phase 1B, Multicentre, Randomized, Double-Blinded, and PLacebo-Controlled Study of the Antiviral Activity, Safety, Tolerability, and PK of Multiple Ascending Doses of VCH-916 in the Treatment Naive or Experienced Subjects With Chronic Hep C-Infection.
Brief Title: Safety,Tolerability and Pharmacokinetics of Multiple Ascending Doses of VCH 916 in Subjects With Chronic Hep C Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: ViroChem Pharma (Industry); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCH 916-103
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-02

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): VCH-916 100 mg three times a day (t.i.d.)
  Interventions: Drug: VCH 916; Drug: Placebo
- Cohort 2 (Experimental): VCH-916 200 mg (t.i.d.)
  Interventions: Drug: VCH 916; Drug: Placebo
- Cohort 3 (Experimental): VCH-916 300 mg twice daily for three days
  Interventions: Drug: VCH 916; Drug: Placebo
- cohort 4 (Experimental): VCH-916 400 mg twice daily for three days
  Interventions: Drug: VCH 916; Drug: Placebo

INTERVENTIONS:
Drug: VCH 916 — Dose escalation study with a full review of all safety data following each cohort.
Drug: Placebo — Dose escalation study with a full review of all safety data following each cohort.

SUMMARY:
The purpose of this study is to determine whether a 3-day course of therapy with orally administered VCH-916 given at different dosages can effectively reduce the amount of circulating virus (i.e., viral load) in patients with early-stage chronic hepatitis C-infection. This study will also evaluate the safety and tolerability of treatment with VCH-916. Blood samples will also be taken to measure the levels of VCH-916 present in plasma at various time points during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 60 years of age
* No evidence of cirrhosis or have liver fibrosis corresponding to Metavir Stages 0 to 3
* Subject's liver disease is stable with ALT values < 5 X ULN
* Serologic evidence of detectable plasma HCV-RNA of ≥ 100,000 IU/ml at screening
* Documented HCV Genotype 1 chronic hepatitis C.
* Judged to be in good health on the basis of medical history and physical examination
* All other hematology and clinical chemistry must be within normal limits or show no clinically significant abnormalities.
* Be treatment-naïve or experienced.
* For female subjects, must not be pregnant or breastfeeding and must be postmenopausal, surgically sterile, abstinent, or using two proven methods of birth control.
* Sexually active male subjects, must be practicing acceptable methods of contraception during the treatment period
* Female subjects of childbearing potential must have a negative serum ß-HCG pregnancy test at screening and a negative urine pregnancy test on Day 1 before the first dose of study drugs.
* Agree not to participate in other clinical trials for the duration of his/her participation in this clinical trial.

Exclusion Criteria:

* Be participating in any other clinical studies or have participated in another clinical trial within the last 30 days before study drug administration, or participation in more than 2 drug studies in the last 12 months (exclusive of the current study).
* Be actively taking hard illicit drugs within 12 months prior to the screening visit or alcohol.
* Have a Child-Pugh score > than 5.
* Have evidence of liver cirrhosis including histological evidence of hepatic cirrhosis on any liver biopsy.
* Have any cause of liver disease other than chronic hepatitis C-infection
* Active or malignant disease or suspicion or history of malignant disease within five previous years (except for adequately treated basal cell carcinoma).
* Have clinically significant electrocardiogram abnormalities and/or cardiovascular dysfunction within the previous 6 months
* Have significant renal, pulmonary, gastrointestinal absorption, or neurological diseases, or neoplasia.
* Have a history of psychiatric disorders determined by the investigator to contraindicate therapy.
* Have uncontrolled Type 1 or Type II diabetes.
* Antinuclear antibody titer ≥1:320.
* Coinfection with hepatitis B and/or HIV 1 or HIV 2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to assess the antiviral activity, safety, and tolerability of VCH-916 monotherapy in adult subjects with chronic HCV-infection. | Day 1 to Day 17 visits

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) profile of VCH-916 in HCV-infected adults. | Day 1 visit
To establish the relationship between VCH-916 plasma levels and corresponding HCV RNA reduction with the administered dosages of VCH-916 in adults. | Day 1 to Day 4 visits
To study the kinetics of plasma HCV RNA following treatment for up to three(3) days with VCH-916. | Day 1 to Day 4 visits

CONTACTS AND LOCATIONS:
Overall Officials: John McHutchison, MD, Principal Investigator — Duke Clinical Research Institute
Locations (5):
- United States (2):
  - The Liver INstitute at Methodist Dallas, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
- Canada (2):
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico